CLINICAL TRIAL: NCT00728247
Title: Objective Kinematic Correlates of Palpatory Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Tamara Reid Bush and Joseph Vorro, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Bush-headneck
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: Cervical Spine
Keywords: Cervical Spine; Kinematics; Manipulation; Biomechanics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Manual Therapy Techniques — One of the following will be selected(1) soft-tissue stretch, (2) myofascial release, (3) muscle energy, or (4) functional (indirect) method

SUMMARY:
Hypothesis: Kinematic parameters can be used to monitor changes in three-dimensional head movements after Manual Therapy treatments.

Subjects who have some level of cervical dysfunction will be examined by an experienced Osteopathic physician. During the clinical assessment of cervical lateral flexion, kinematic data will be recorded. Subjects will be treated using manual therapy techniques and kinematic data will be recorded again at set intervals after the treatment.

DETAILED DESCRIPTION:
The physician providing treatment will use, depending on his professional judgment for each subject, one of four treatment modalities: (1) soft-tissue stretch, (2) myofascial release, (3) muscle energy, or (4) functional (indirect) method. These modalities are standard to the care and practice of osteopathic manual medicine, they are taught in the Osteopathic curriculum, and they are practiced each day at the Michigan State University Clinical Center.

After the initial treatment, there will be an immediate follow-up kinematic test to collect the 3-D motion data. Then, subjects will return for subsequent kinematic assessments at: 24 hours post treatment, 48 hours post treatment and seven days post treatment. At the seven day mark, subjects will be evaluated as in the initial assessment and the physician will use his professional judgment to determine if the subject would benefit from a second treatment. If so, then the process of treatment and kinematic assessment would occur a second time, with kinematic assessment 24 hours post treatment, 48 hours post treatment and seven days post treatment. A maximum of two treatment sessions will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females over the age of 18 and up to 100 years of age

Exclusion Criteria:

* Pregnant women and minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Three-dimensional kinematics | Same day, 24 hours, 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Biomechanical Design Research Laboratory, East Lansing, Michigan, United States